CLINICAL TRIAL: NCT04522219
Title: Contribution of Contrast Enhanced Ultrasound in the Diagnosis of Adnexal Torsion: a Prospective Comparative Study
Brief Title: Contribution of Contrast Enhanced Ultrasound in the Diagnosis of Adnexal Torsion
Acronym: AGATA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulties in recruiting patients
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERTHOLDT Charline, Principal investigator (Obstetrician, Medical Doctor), Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-000993-27
Record Dates: First submitted 2020-07-21; First posted 2020-08-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Adnexal Torsion
Keywords: adnexal; torsion; ovarian; contrast enhanced ultrasound
MeSH Terms: conditions — Ovarian Torsion

STUDY DESIGN:
Intervention Model Description: Phase 3b, prospective, Case-Control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): Diagnosis of adnexal torsion confirmed by the surgical intervention: woman allocated to case group
  Interventions: Diagnostic Test: Contrast enhanced ultrasound
- Control group (Experimental): Diagnosis of adnexal torsion not confirmed by the surgical intervention: woman allocated to control group
  Interventions: Diagnostic Test: Contrast enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast enhanced ultrasound — Acquisition of contrast enhanced ultrasound. Contrast agent: SonoVue®: Hexafluoride (SonoVue®, injectable solution to solubilisate, 8µg/mL) is injected in all patients

SUMMARY:
Clinical diagnosis of adnexal torsion is difficult because the symptomatology is dominated by abrupt onset pelvic pain, an aspecific sign which does not allow a diagnosis of certainty to be made.

To confirm the diagnosis, the reference examination is pelvic ultrasound with Doppler flow analysis. However, its intake is low, its sensitivity varies from 46 to 73% depending on the studies. Other imaging techniques have been considered, such as MRI, with a sensitivity far superior to ultrasound, but its difficult accessibility, in particular in the context of an emergency, makes it unusable in clinical practice.

The use of ultrasound with the injection of an ultrasound contrast agent, strict intravascular, seems to be an interesting technique to assess the perfusion parameters of the ovary and improve the diagnostic sensitivity of the adnexal torsion. Its interest has already been demonstrated in the diagnosis of testicular torsion in animals but to date, no study has evaluated its contribution in adnexal torsion.

DETAILED DESCRIPTION:
The primary objective is to evaluate the diagnostic performance of contrast enhanced ultrasound for the diagnosis of adnexal torsion in women with suspected adnexal torsion.

The secondary objectives are:

1. To describe the perfusion parameters of the ovaries by contrast enhanced ultrasound
2. To compare performance diagnosis of contrast ultrasound and bidimensional Doppler for the detection of adnexal torsion.
3. To describe the perfusion parameters of the ovarian as a function of the degree of adnexal torsion.
4. To compare perfusion parameters before and after ovarian detorsion
5. To describe perfusion parameters of the ovarian by using MicroVascular Flow technique
6. To assess the contribution of qualitative contrast ultrasound for the diagnosis of adnexal torsion (without clinical context)
7. To assess inter-observer agreement on the qualitative analysis of ultrasound, without clinical context and then with clinical context.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years old
* Woman affiliated to a social security
* Woman having received complete information on the organization of the research and having given her informed consent in written form.
* Planned surgical intervention for suspected adnexal torsion

Exclusion Criteria:

* Patients under a measure of legal protection,
* Contraindication to contrast injection Hypersensitivity to sulfur hexafluoride or any of the other ingredients, history of cardiac disease, respiratory distress syndrome, severe pulmonary hypertension..

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Signal intensity measurement | through study completion, on average of 36 months
  to assess sensitivity, specificity, positive and negative predictive value of contrast enhanced ultrasound for detection of adnexal torsion in women with suspected adnexal torsion with realization of ROC curves

SECONDARY OUTCOMES:
vascularization of the ovaries on contrast enhanced ultrasound. | through study completion, an average of 36 months
  Measurement of perfusion parameters of the suspected ovarian torsion and the contralateral ovary if available:
diagnostics performance | through study completion, an average of 36 months
  Measurement of signal intensities to assess sensibility and specificity of contrast enhanced ultrasound and bidimensional (2D) Doppler.
vascularization of the ovaries according to the degree of torsion | through study completion, an average of 36 months
  Comparison of perfusion parameters of the ovary with the degree of torsion. The degree of torsion is defined by the number of twists (number of turns around the axis) detected during the surgical procedure.
vascularization of the ovaries before and after detorsion | through study completion, an average of 36 months
  Measurement of signal intensities before and after ovarian detorsion
Micro Vascular Flow technique | through study completion, an average of 36 months
  Measurement of signal intensities obtained by Micro Vascular Flow technique
Qualitative evaluation of contrast enhancement | through study completion, an average of 36 months
  Presence or absence of contrast within the ovary. The presence of torsion is defined as for the primary objective.
Reproducibility of qualitative evaluation of contrast enhancement | through study completion, an average of 36 months
  Diagnosis of adnexal torsion assessed by two observer on qualitative contrast ultrasound, without and with clinical context. Concordance will be assessed by the kappa coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Charline BERTHOLDT, Study Chair — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pillot R, Hossu G, Cherifi A, Guillez K, Morel O, Beaumont M, Fijean AL, Bertholdt C. Contribution of contrast-enhanced ultrasound in the diagnosis of adnexal torsion (AGATA): protocol for a prospective comparative study. BMJ Open. 2023 Aug 24;13(8):e073301. doi: 10.1136/bmjopen-2023-073301. PMID 37620263